CLINICAL TRIAL: NCT00989664
Title: Multicenter, Pivotal Phase III Study of Iodine-131 Anti-B1 Antibody (Murine) Radioimmunotherapy for Chemotherapy Refractory Low Grade B Cell Lymphomas and Low Grade Lymphomas That Have Transformed to Higher Grade Histologies
Brief Title: Pivotal Study of Iodine I 131 Tositumomab for Chemotherapy-refractory Low-grade or Transformed Low-grade B-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104504
Expanded Access: Available
Record Dates: First submitted 2009-10-01; First posted 2009-10-05 (Estimated); Results first posted 2012-04-10 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-10

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: non-Hodgkin's Lymphoma; radioimmunotherapy; NHL; Bexxar; lymphoma; Tositumomab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — tositumomab I-131

ARMS (1):
- open-label single arm (Experimental): Tositumomab and Iodine-131 Tositumomab radioimmunotherapy for chemotherapy-refractory low-grade B-cell lymphomas and low-grade lymphomas that have transformed to higher grade histologies.
  Interventions: Biological: Tositumomab and Iodine I 131 Tositumomab

INTERVENTIONS:
Biological: Tositumomab and Iodine I 131 Tositumomab — Dosimetric Dose: 450 mg of TST infused over 70 minutes (inclusive of a 10-minute flush) immediately followed by I-131 TST (35 mg of TST, of which 1-2 mg had been labeled with 5 mCi of Iodine-131) infused over 30 minutes (inclusive of a 10-minute flush).
  Therapeutic Dose: 7 to 14 days after the dosimetric dose, 450 mg of TST infused over 70 minutes (inclusive of a 10-minute flush) immediately followed by I-131 TST (35 mg of TST labeled with enough Iodine-131 to administer the specified whole body radiation dose determined for the subject) infused over 30 minutes (inclusive of a 10-minute flush). The desired total body dose was 65 cGy for subjects with a baseline platelet count of 100,001-149,999/mm3 and 75 cGy for patients with a baseline platelet count ≥150,000/mm3. Obese patients received an attenuated dose by not including subject mass over 137% of their calculated lean body mass in their calculated lean body mass in the dose calculation.

SUMMARY:
The results from Phase 1/2 (RIT-I-000) and Phase 2 (RIT-II-001) studies of Tositumomab and Iodine I 131 Tositumomab (TST/I-131 TST) demonstrated that TST/ I-131 TST produced a high response rate in patients with chemotherapy-relapsed/refractory, low-grade or transformed low-grade Non-Hodgkin's Lymphoma (NHL). On the basis of these results this study was designed to compare the efficacy of TST/ I-131 TST to the last qualifying chemotherapy regimen in patients with chemotherapy-refractory, low-grade or transformed low-grade NHL.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥18 years of age with histologically confirmed at initial diagnosis, previously treated (at least 2 prior chemotherapy regimens), low-grade NHL or low-grade lymphoma that had transformed to intermediate- or high-grade histology.

Exclusion Criteria:

* Subjects with more than an average of 25% of the intratrabecular marrow space involved by lymphoma in bone marrow biopsy specimens as assessed microscopically within 42 days of study entry. Bilateral posterior iliac crest core biopsies are required if the percentage of intratrebecular space involved exceeds 10% in a unilateral biopsy. The mean of bilateral biopsies must be no more than 25%.
* Cytotoxic chemotherapy, radiation therapy, immunosuppressants, or cytokine treatment within 4 weeks prior to study entry or persistent clinical evidence of toxicity.
* Prior stem cell transplant.
* Active obstructive hydronephrosis.
* Evidence of active infection requiring intravenous (IV) antibiotics at the time of study entry.
* New York Heart Association Class III or IV heart disease or other serious illness that would preclude evaluation.
* Prior malignancy other than lymphoma, except for adequately treated skin cancer, in situ cervical cancer, or other cancer for which the subject has been disease-free for 5 years.
* Known HIV infection.
* Known brain or leptomeningeal metastases.
* Subjects who are pregnant or nursing.
* Previous allergic reactions to iodine. This does not include reactions to intravenous iodine-containing contrast materials.
* Prior exposure to monoclonal or polyclonal antibodies of any non-human species for either diagnostic or therapeutic purposes, including engineered chimeric and humanized antibodies.
* Prior radioimmunotherapy.
* Progressive disease within 1 year of irradiation arising in a field that has been previously irradiated with >3500 cGy.
* Current use of either approved or non-approved (through another protocol) anti-cancer drugs or biologics
* De novo intermediate- or high-grade lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 1996-11; Primary Completion 2004-01 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kaminski MS, Zelenetz AD, Press OW, Saleh M, Leonard J, Fehrenbacher L, Lister TA, Stagg RJ, Tidmarsh GF, Kroll S, Wahl RL, Knox SJ, Vose JM. Pivotal study of iodine I 131 tositumomab for chemotherapy-refractory low-grade or transformed low-grade B-cell non-Hodgkin's lymphomas. J Clin Oncol. 2001 Oct 1;19(19):3918-28. doi: 10.1200/JCO.2001.19.19.3918. PMID 11579112
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 104504 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104504 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104504 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104504 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104504 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104504 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104504 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) received radioimmunotherapy of tositumomab (TST) and Iodine I 131 TST in 2 phases (Ph.): Ph. 1, dosimetric dose; Ph. 2, therapeutic dose. Par. were evaluated until disease progression, they died, or they were on study for 2 years. Par. completing 2 years of study could enter a long-term follow-up study (BEX104526; NCT00240591).
Groups:
- TST and I 131 TST: Participants received a dosimetric dose (DD) consisting of 450 milligrams (mg) of tositumomab (TST) intravenously (IV) immediately followed by I 131 TST (35 mg of TST, of which 1-2 mg was labelled with 5 millicurie [mCi] of I 131) IV. The therapeutic dose (TD) consisted of 450 mg of TST IV, immediately followed by a participant-specific dose of I 131 TST (35 mg of TST labelled with I 131 to administer 75 centigray [cGy] or 65 cGy). The TD was administered 7-14 days after the DD. Participants who had completed at least 2 years of follow up after administration of TST/I 131 TST during the TD phase and had signed the informed consent to participate in the Long-Term Follow-Up (LTFU) study (BEX104526) were followed for up to 10 years. Participants did not receive any study medication during the LTFU study.
Period: Dosimetric and Therapeutic Treatment
Arm/Group | TST and I 131 TST
Started | 61
Completed | 0
Not Completed | 61
Not completed — Non-compliant or Uncooperative | 1
Not completed — Condition/Illness; Study Drug Unrelated | 2
Not completed — Progressive Disease | 49
Not completed — Death | 1
Not completed — Enrolled into Study BEX104526 | 7
Not completed — Did Not Receive Study Drug | 1
Period: Long-Term Follow-Up
Arm/Group | TST and I 131 TST
Started | 14 (14 of the 61 participants withdrawing from Study BEX104504 enrolled in the LTFU study.)
Completed | 11
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics are summarized for the Intent-to-Treat (ITT) Exposed Population, comprised of all participants who were enrolled in the study and received at least one dose of study drug.
  Years | 59.4 (10.5)
Gender [Count of Participants; unit: Participants] — Baseline characteristics are summarized for the Intent-to-Treat (ITT) Exposed Population, comprised of all participants who were enrolled in the study and received at least one dose of study drug.
  Participants
    Female | 22
    Male | 38
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics are summarized for the ITT Exposed Population, comprised of all participants who were enrolled in the study and received at least one dose of study drug.
  participants
    White | 58
    Hispanic | 1
    Black | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Par.) Receiving TST and I 131 TST With a Response >=30 Days Versus Par. With a Response >=30 Days After Their Last Qualifying Chemotherapy Regimen (LQCR), Masked Independent Randomized Radiology and Oncology Review (MIRROR) Panel
Description: Par. with response are those with complete response (CR; complete resolution of all disease-related radiological abnormalities and the disappearance of all signs/symptoms related to disease), complete response unconfirmed (CRu; meets characteristics of CR, except the nodal size hasn't regressed sufficiently, or there is indeterminate bone marrow), or partial response (PR; >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions with no new lesions). Participants' LQCR was used as a comparator for subsequent treatment with Iodine I 131TST.
Time Frame: Participants were evaluated for up to 99.1 months in Study 104504 or were followed in the long-term follow-up study for up to 141.5 months
Population: ITT Exposed Population
Measure: Number; unit: participants
Groups:
- LQCR: Participants previously treated with at least two chemotherapy regimes before enrolling in Study BEX104504
Arm/Group | TST and I 131 TST | LQCR
Number analyzed (Participants) | 60 | 60
participants | 26 | 5
Statistical Analysis 1: Comparison: TST and I 131 TST vs LQCR; Test type: Superiority or Other; p < 0.001, McNemar

2. Primary Outcome: Duration of Response for Par. Receiving TST and I 131 TST With a Response >=30 Days Versus the Number of Par. With a Response >=30 Days After Their LQCR, as Assessed by the MIRROR Panel
Description: Duration of response is defined as the time from the first documented response (for par. with complete response, complete response unconfirmed, or partial response) until disease progression (DP). DP is defined as a >=25% increase from the nadir value (lowest laboratory value recorded following administration of the study medication) of the sum of the products of the longest perpendicular diameters of all measurable lesions or the appearance of any new lesion. Individual lesions must be >2 centimeters (cm) in diameter by radiographic evaluation or >1 cm in diameter by physical examination.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants with complete response, complete response unconfirmed, or partial response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and I 131 TST | LQCR
Number analyzed (Participants) | 33 | 17
months | 6.5 [3.1 to 11.3] | 3.5 [2.5 to 4.5]

3. Secondary Outcome: Number of Participants With Any Uncofirmed Response (CR, Clinical Complete Response [CCR], or PR), CR, CCR, CR+CCR, and PR), as Assessed by the Investigator
Description: Participants with response include those with CR, CCR, or PR. Criteria for CR: complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease. Criteria for CCR: complete resolution of all disease-related symptoms, but residual foci, thought to be residual scar tissue, are present. Criteria for PR: >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions with no new lesions.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants evaluable for response were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 59
participants
  Response (CR, CCR, or PR) | 39
  CR | 11
  CCR | 1
  CR+CCR | 12
  PR | 27

4. Secondary Outcome: Number of Participants With Any Confirmed Response (CR, CCR, or PR), Confirmed CR, Confirmed CCR, Confirmed CR+CCR, and Confirmed PR, as Assessed by Investigator
Description: Responses had to be confirmed by 2 separate evaluations occurring >=4 weeks apart. Par. with confirmed response include those with CR, CCR , or PR. A confirmed response (CR/CCR/PR) had to be confirmed by a consecutive response (>=28 days [ 4 weeks] later) that was the same or better. Individual confirmed response data only counts that response confirmed by the same response; thus, not all possible combinations are represented.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants evaluable for confirmed response were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 50
participants
  Confirmed Response (CR, CCR, or PR) | 30
  CR | 9
  CCR | 1
  CR+CCR | 11
  PR | 18

5. Secondary Outcome: Time to Progression of Disease or Death, as Assessed by the Investigator
Description: Time to progression or progression-free survival is defined as the time from the dosimetric dose to the first documented occurrence of disease progression or death. Disease progression is defined as a >=25% increase from the nadir value (lowest laboratory value recorded following administration of the study medication) of the sum of the products of the longest perpendicular diameters of all measurable lesions or the appearance of any new lesion. Individual lesions must be >2 cm in diameter by radiographic evaluation or >1 cm in diameter by physical examination.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants who experienced disease progression or died were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 54
months | 4.7 [3.3 to 5.8]

6. Secondary Outcome: Time to Treatment Failure, as Assessed by the Investigator
Description: Time to treatment failure is defined as the length of time from the date of enrollment to the first incidence of treatment withdrawal, study removal, progression, and/or alternative therapy for the participant's lymphoma, or death.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants who experienced treatment failure were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 54
months | 4.6 [3.2 to 5.8]

7. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the treatment start date to the date of death from any cause.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants who died during the study and during the follow-up period were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 48
months | 30.1 [17.1 to 39.9]

8. Secondary Outcome: Number of Participants With Responses of CR, CCR, CR+CCR, and PR Following TST and I 131 TST and Following the LQCR, as Assessed by the Investigator
Description: as for outcome 3
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants evaluable for response were analyzed.
Measure: Number; unit: participants
Groups:
- LQCR: Participants treated with at least two chemotherapy regimens before enrolling in study BEX104504
Arm/Group | TST and I 131 TST | LQCR
Number analyzed (Participants) | 59 | 60
participants
  Response (CR, CCR, or PR) | 39 | 17
  CR | 11 | 1
  CCR | 1 | 1
  CR+CCR | 12 | 2
  PR | 27 | 15

9. Secondary Outcome: Number of Participants With the Indicated Adverse Events (AE) Related to Study Drug Experienced by at Least 5% of Participants
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The Investigator assessed whether the adverse event was related to study drug.
Time Frame: as for outcome 1
Population: ITT Exposed Population. All participants who experienced any AE related to study drug were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 57
participants
  Absolute Neutrophil Count (ANC) <1000 cells/cm^3 | 35
  Platelets <50000 cells/cm^3 | 29
  White Blood Cells (WBC) <2000 cells/cm^3 | 29
  Hemoglobin <8.0 grams/deciliter (g/dL) | 13
  Fatigue | 27
  Pyrexia | 19
  Chills | 11
  Nausea | 16
  Vomiting | 9
  Diarrhoea | 4
  Thrombocytopenia | 10
  Neutropenia | 9
  Anaemia | 7
  Leukopenia | 4
  Pruritus | 8
  Rash | 4
  Night sweats | 3
  Cough | 7
  Dyspnoea | 7
  Throat irritation | 4
  Productive cough | 3
  Headache | 5
  Dizziness | 3
  Somnolence | 3
  Decreased appetite | 11
  Arthralgia | 5
  Myalgia | 5
  Pain in extremity | 3
  Myelodysplastic syndrome | 4
  Hypothyroidism | 7
  Hypotension | 5
  Tachycardia | 3

10. Secondary Outcome: Number of Participants With the Indicated Grade 3 or Grade 4 AEs Experienced by at Least 5% of Participants
Description: AEs were graded using the Common Toxicity Criteria from the Cancer Therapy Evaluation Program, Division of Cancer Therapy, National Cancer Institute. Grades: 0 = No AE or within normal limits; 1 = Mild AE; 2 = Moderate AE; 3 = Severe and undesirable AE; 4 = Life-threatening or disabling AE; 5 = Death related to AE.
Time Frame: as for outcome 1
Population: ITT Exposed Population. All participants who experienced Grade 3 or Grade 4 AEs were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 51
participants
  ANC <1000 cells/cm^3 | 35
  Platelets <50000 cells/cm^3 | 29
  WBC <2000 cells/cm^3 | 29
  Hemoglobin <8.0 g/dL | 13
  Myelodysplastic syndrome | 4
  Neutropenia | 9
  Thrombocytopenia | 8
  Anaemia | 4
  Leukopenia | 3
  Dyspnoea | 3
  Pleural effusion | 3

11. Secondary Outcome: Number of Participants With the Indicated Grade 3 or Grade 4 AEs Related to Study Drug and Experienced by at Least 5% of Participants
Description: AEs were graded using the Common Toxicity Criteria from the Cancer Therapy Evaluation Program, Division of Cancer Therapy, National Cancer Institute. Grades: 0 = No AE or within normal limits; 1 = Mild AE; 2 = Moderate AE; 3 = Severe and undesirable AE; 4 = Life-threatening or disabling AE; 5 = Death related to AE. The Investigator assessed whether the AE was possibly or probably related to study drug. In addition, all laboratory-derived hematologic toxicities (values outside the normal range) were assumed to be possibly or probably related to study drug.
Time Frame: as for outcome 1
Population: ITT Exposed Population. All participants who experienced Grade 3 or 4 AEs related to study drug were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 46
participants
  ANC <1000 cells/cm^3 | 35
  Platelets <50000 cells/cm^3 | 29
  WBC <2000 cells/cm^3 | 29
  Hemoglobin <8.0 g/dL | 13
  Neutropenia | 9
  Thrombocytopenia | 8
  Anaemia | 4
  Leukopenia | 3
  Myelodysplastic syndrome | 4

12. Secondary Outcome: Number of Participants With the Indicated Primary Cause of Death
Description: The primary cause of death of the participants was assessed by the Investigator.
Time Frame: as for outcome 1
Population: ITT Exposed Population. All participants who died during the study were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 48
participants
  Progression of lymphoma | 37
  Complications related to study drug | 0
  Other | 11

13. Secondary Outcome: Number of Participants With the Indicated Time to Death From the Last Dose of Study Drug
Description: Time to death from the last dose of study drug is the time period difference between when study drug treatment stopped and when death occurred.
Time Frame: as for outcome 1
Population: ITT Exposed Population. All participants who died during the study were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 48
participants
  <=30 Days | 1
  >30 Days | 47

14. Secondary Outcome: Number of Participants With the Indicated Fatal Serious Adverse Events (SAE) Unrelated to Study Drug
Description: An SAE is any event occurring at any dose that results in any of the following: death, a life-threatening adverse drug experience (ADE; at immediate risk of death from the experience as it occurred), inpatient hospitalization/prolongation of existing hospitalization, a persistent/significant disability/incapacity, or a congenital anomaly/birth defect. Medical events that may not result in death, be life threatening, or require hospitalization may be considered to be a serious ADEs when based upon appropriate medical judgment. Relatedness was based on the Investigator's medical judgment.
Time Frame: as for outcome 1
Population: ITT Exposed Population. All participants who experienced fatal SAEs were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 10
participants
  Pneumonia aspiration | 1
  Non-Hodgkins lymphoma | 2
  Encephalopathy | 1
  Dyspnea | 1

15. Secondary Outcome: Number of Participants With the Indicated Fatal SAEs Related to Study Drug
Description: An SAE is any event occurring at any dose that results in any of the following: death, a life-threatening adverse drug experience (ADE; at immediate risk of death from the experience as it occurred), inpatient hospitalization/prolongation of existing hospitalization, a persistent/significant disability/incapacity, or a congenital anomaly/birth defect. Medical events that may not result in death, be life threatening, or require hospitalization may be considered to be a serious AEs when based upon appropriate medical judgment. Relatedness was based on the Investigator's medical judgement.
Time Frame: as for outcome 1
Population: ITT Exposed Population. All participants who experienced fatal SAEs were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 10
participants
  Lung adenocarcinoma | 1
  Myelodysplastic syndrome | 2
  Encephalopathy | 1
  Pulmonary hemorrhage | 1

16. Secondary Outcome: Number of Participants With the Indicated SAEs Related to Study Drug
Description: An SAE is any event occurring at any dose that results in any of the following: death, a life-threatening adverse drug experience (ADE; at immediate risk of death from the experience as it occurred), inpatient hospitalization/prolongation of existing hospitalization, a persistent/significant disability/incapacity, or a congenital anomaly/birth defect. Medical events that may not result in death, be life threatening, or require hospitalization may be considered to be a serious ADEs when based upon appropriate medical judgment. Relatedness was based on the Investigator's medical judgement.
Time Frame: as for outcome 1
Population: ITT Exposed Population. All participants who experienced SAEs were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 19
participants
  Myelodysplastic syndrome | 4
  Squamous cell carcinoma | 2
  Basal cell carcinoma | 1
  Colon cancer stage 0 | 1
  Lung adenocarcinoma | 1
  Refractory anaemia with an excess of blasts | 1
  Squamous cell carcinoma of skin | 1
  Anaemia | 2
  Leukopenia | 1
  Neutropenia | 1
  Chronic obstructive pulmonary disease | 1
  Dyspnoea | 1
  Pulmonary haemorrhage | 1
  Pneumocystis jiroveci pneumonia | 1
  Pneumonia | 1
  Atrial flutter | 1
  Subdural haematoma | 1
  Arthralgia | 1
  Encephalopathy | 1

17. Secondary Outcome: Number of Participants With the Indicated Type of Infection
Description: An infection is the colonization of a host organism by a parasite species. Infecting parasites seek to use the host's resources to reproduce, often resulting in disease. Specimen samples of the body fluid are cultured for testing whether the infectious organism is present and grown in the culture media to assess the growth pattern of the organisms present in the specimen. The culture results could be positive or negative. The positive culture results indicate that the tested participant has the infection under investigation, in which case therapeutic treatment with anti-infective is required.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants who experienced any infection were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 59
participants
  Any Infection; n=59 | 15
  No Infection; n=59 | 44
  Sepsis; n=15 | 0
  Pneumonia; n=15 | 5
  Other Infections; n=15 | 14

18. Secondary Outcome: Number of Participants With an Infection for Which Anti-infectives Were Administered
Description: Anti-infectives are capable of acting against infection, by inhibiting the spread of an infectious agent or by killing the infectious agent outright. Anti-infective is a general term that encompasses antibacterials, antibiotics, antifungals, antiprotozoans, and antivirals.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants who had an infection during the study and during the follow-up period were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 15
participants
  Anti-infective Administered | 12
  Anti-infective Not Administered | 3

19. Secondary Outcome: Number of Participants Who Were Negative for Human Anti-murine Antibodies (HAMA) at Baseline (Before Receiving the Dosimetric Dose) But Positive or Negative After Receiving the Dosimetric Dose
Description: The administration of murine antibodies may form HAMA. A HAMA assay was performed using the ImmunoSTRIP HAMA IgG enzyme-linked immune absorbent assay by a central laboratory (Covance Classic Laboratory Services, Indianapolis, IN). Fludarabine, a known immunosuppressant, might decrease HAMA production in addition to reducing bone marrow involvement. To be "positive," a participant had to have a positive HAMA assessment at any follow-up visit.
Time Frame: HAMA was measured at baseline; Day5; Weeks 7, 17, 25; and then every 12 months while in study BEX104526. Participants were evaluated for up to 99.1 months in Study 104504 or were followed in the long-term follow-up study for up to 141.5 months
Population: ITT Exposed Population. Only those participants evaluable for HAMA were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 58
participants
  Positive | 5
  Negative | 53

20. Secondary Outcome: Time to HAMA Positivity From the First Dosimetric Dose
Description: HAMA are human immunoglobulins with specificity for mouse immunoglobulins. HAMA assays were conducted in the laboratory to measure conversion to HAMA positivity following treatment. Time to HAMA positivity was calculated as the difference between the day on which HAMA positivity occurred and the first dosimetric dose administration day.
Time Frame: as for outcome 19
Population: ITT Exposed Population. Participants who converted from being negative for HAMA at Baseline to being positive for HAMA following treatment were analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 5
days | 279 [21 to 426]

21. Secondary Outcome: Number of Participants With the Indicated Grade 3 or Grade 4 Hematologic Toxicities
Description: Adverse events were graded using the Common Toxicity Criteria from the Cancer Therapy Evaluation Program, Division of Cancer Therapy, National Cancer Institute. Grades: 0 = No adverse event or within normal limits; 1 = Mild adverse event; 2 = Moderate adverse event; 3 = Severe and undesirable adverse event; 4 = Life-threatening or disabling adverse event; 5 = Death related to adverse event. Grade 3/4 hematological toxicities: hemoglobin <8.0 g/dL; platelets <50,000 cells per millimeters (mm)^3; ANC <1000 cells per mm^3; WBC <2000 cells per mm^3.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Number; unit: participants
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 60
participants
  ANC | 35
  Hemoglobin | 13
  Platelets | 29
  WBC count | 29

22. Secondary Outcome: Number of Participants With Hypothyroidism Prior to Therapy and After the Therapeutic Dose
Description: Thyroid function was determined periodically, including during follow-up, in order to assess if there was any effect of the Iodine 131 on thyroid function. Hypothyroidism is a condition in which the thyroid gland does not make enough thyroid hormone.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Participants who were evaluable for thyroid function assessment were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and I 131 TST
Number analyzed (Participants) | 52
participants
  Prior to therapy | 8
  After therapeutic dose | 7

ADVERSE EVENTS:
Time Frame: Participants were evaluated until death or were followed in the long-term follow-up study for up to 10 years.
Arm/Group | TST and I 131 TST
Serious Adverse Events (participants affected / at risk) | 30/60
Other Adverse Events (participants affected / at risk) | 59/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TST and I 131 TST (N=60)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Refractory anaemia with an excess of blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Superior vena caval occlusion (Vascular disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardiomegaly (Cardiac disorders) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Encephalopathy (Nervous system disorders) | 2
Nephropathy (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Hypercalcaemia of malignancy (Endocrine disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TST and I 131 TST (N=60)
Fatigue (General disorders) | 29
Pyrexia (General disorders) | 22
Chills (General disorders) | 11
Asthenia (General disorders) | 6
Oedema peripheral (General disorders) | 6
Chest pain (General disorders) | 4
Pain (General disorders) | 3
Chest discomfort (General disorders) | 2
Oedema (General disorders) | 2
Early satiety (General disorders) | 1
Feeling cold (General disorders) | 1
Feeling jittery (General disorders) | 1
Hunger (General disorders) | 1
Infusion site extravasation (General disorders) | 1
Malaise (General disorders) | 1
Nodule (General disorders) | 1
Swelling (General disorders) | 1
ANC < 1,000 cells/mm^3 (Investigations) | 35
Platelets <50000 cells/mm^3 (Investigations) | 29
WBC < 2000 cells/mm^3 (Investigations) | 29
Hemoglobin < 8.0 g/dL (Investigations) | 13
Nausea (Gastrointestinal disorders) | 21
Diarrhoea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 12
Abdominal pain (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 5
Abdominal discomfort (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Diverticulum (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Tongue ulceration (Gastrointestinal disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Bone lesion (Musculoskeletal and connective tissue disorders) | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia exertional (Respiratory, thoracic and mediastinal disorders) | 1
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8
Night sweats (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 5
Bronchitis (Infections and infestations) | 4
Herpes zoster (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 3
Oral herpes (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Haemophilus infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Keratitis herpetic (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 7
Somnolence (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 4
Amnesia (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Mental impairment (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Peroneal nerve palsy (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Neutropenia (Blood and lymphatic system disorders) | 8
Anaemia (Blood and lymphatic system disorders) | 6
Leukopenia (Blood and lymphatic system disorders) | 3
Lymph node pain (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Lymphatic disorder (Blood and lymphatic system disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 15
Dehydration (Metabolism and nutrition disorders) | 1
Folate deficiency (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 6
Deep vein thrombosis (Vascular disorders) | 2
Flushing (Vascular disorders) | 2
Aortic stenosis (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Weight decreased (Investigations) | 4
Blood pressure decreased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Heart sounds abnormal (Investigations) | 1
Occult blood positive (Investigations) | 1
Respiratory rate increased (Investigations) | 1
Weight increased (Investigations) | 1
Depression (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Boredom (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Tearfulness (Psychiatric disorders) | 1
Tachycardia (Cardiac disorders) | 6
Palpitations (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 7
Upper limb fracture (Injury, poisoning and procedural complications) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
Conjunctivitis (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye oedema (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Ear pain (Ear and labyrinth disorders) | 1
Multiple allergies (Immune system disorders) | 1
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast pain (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.